CLINICAL TRIAL: NCT07003464
Title: Efficacy and Safety of Zanubrutinib, Obinutuzumab, and Bendamustine (ZGB) Regimen for First-Line Treatment of Chronic Lymphocytic Leukemia: A Single-Arm, Prospective Study
Brief Title: Phase II Trial of Zanubrutinib, Obinutuzumab, Bendamustine (ZGB) as First-Line Therapy for Chronic Lymphocytic Leukemia: A Single-Center Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ou Bai, MD/PHD, Director, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-2024-ZGB-01
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; obinutuzumab; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: This trial follows a single-arm, two-stage, MRD-adapted design to assess both safety and preliminary efficacy of the ZGB regimen.
  Structure: Sequential Two-Stage Intervention Induction Phase (Cycles 1-4): All participants receive Zanubrutinib + Obinutuzumab + Bendamustine (ZGB).
  Consolidation Phase (Cycles 5-6): Only participants achieving peripheral blood uMRD (<0.01% by flow cytometry) after Cycle 4 receive Zanubrutinib + Obinutuzumab (ZG); others discontinue treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZGB arm (Experimental): Single-arm, two-stage, MRD-adapted design to assess both safety and preliminary efficacy of the ZGB regimen.
  Structure: Sequential Two-Stage Intervention： Induction Phase (Cycles 1-4): All participants receive Zanubrutinib + Obinutuzumab + Bendamustine (ZGB).
  Consolidation Phase (Cycles 5-6): Only participants achieving peripheral blood uMRD (<0.01% by flow cytometry) after Cycle 4 receive Zanubrutinib + Obinutuzumab (ZG); others discontinue treatment.
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg (2 tablets) BID. Each 4-week period constitutes one treatment cycle.
Drug: Obinutuzumab — 1000 mg IV (Days 1, 8, 15 of Cycle 1; Day 1 thereafter).Each 4-week period constitutes one treatment cycle.
Drug: Bendamustine — 70 mg/m² (Days 1-2 per cycle) for induction only (Cycles 1-4).Each 4-week period constitutes one treatment cycle.

SUMMARY:
This is a single arm, open label, national multicenter clinical study included patients with chronic lymphocytic leukemia (CLL). The treatment combines three medications: Zanubrutinib , Obinutuzumab and Bendamustine . Together, these drugs aim to achieve deep remission (no detectable cancer cells) and allow a shorter treatment duration compared to lifelong therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Demographics: Age ≥18 years, regardless of gender.
2. Diagnosis: Confirmed diagnosis of untreated chronic lymphocytic leukemia (CLL) per iwCLL 2018 criteria.
3. Treatment Naivety:

   * No prior systemic therapy for CLL, including:
   * CHOP/COP-based chemotherapy.
   * Regimens containing fludarabine or bendamustine.
   * Anti-CD20 monoclonal antibodies (e.g., rituximab) or BTK inhibitors (e.g., ibrutinib).
   * Chlorambucil or cyclophosphamide (>3 weeks of use).
   * Interferon therapy (>6 months of use).
4. Treatment Indications:

   * Must meet ≥1 of the following (iwCLL 2018 criteria):
   * Hemoglobin <100 g/L (non-hemolytic).
   * Platelets <100×10⁹/L with progressive decline.
   * Lymphadenopathy (longest diameter >10 cm) or massive splenomegaly (>6 cm below costal margin).
   * Constitutional symptoms: unexplained fever (>38°C ×2 weeks), night sweats, or >10% weight loss in 6 months.
   * Rapid disease progression (lymphocyte doubling time <6 months, 50% lymph node growth in 2 months, or rapid cytopenia).
5. Performance Status: ECOG performance status ≤2.
6. Organ Function (within 7 days before enrollment):

   Hematologic:
   * ANC ≥1.0×10⁹/L (without growth factor support).
   * Platelets ≥50×10⁹/L (without transfusion).
   * Hepatic: AST/ALT ≤2.5×ULN; total bilirubin ≤1.5×ULN.
   * Renal: Estimated CrCl ≥30 mL/min (Cockcroft-Gault formula).
7. Consent: Signed informed consent.

Exclusion Criteria:

1. Malignancy: History of active malignancy (excluding CLL) within the past year, including CNS lymphoma.
2. Disease Transformation: Richter transformation or prolymphocytic leukemia (PLL).
3. Autoimmune Cytopenias: Active autoimmune hemolysis or thrombocytopenia requiring corticosteroids.
4. Organ Dysfunction: ALT/AST >3×ULN; total bilirubin >2×ULN; creatinine >1.5×ULN.
5. Comorbidities: Uncontrolled diabetes, cardiac/pulmonary disease, or conditions deemed by investigators to affect study safety.
6. Infections: Active systemic infection requiring IV antibiotics.
7. Bleeding Risks: History of life-threatening hemorrhage or need for high-dose anticoagulation.
8. Recent Surgery: Major surgery within 30 days.
9. Reproductive Status: Pregnancy, lactation, or unwillingness to use contraception.
10. Drug Tolerance: Hypersensitivity to any study drug components.
11. Viral Infections: Active HBV (HBsAg+ or HBV-DNA+) or HCV.
12. Other: Investigator-determined ineligibility (e.g., poor compliance, psychiatric disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Undetectable Minimal Residual Disease (uMRD) Rate | Assessed at the end of Cycle 6 (each cycle = 28 days).
  Proportion of participants achieving uMRD (defined as <1 CLL cell per 10,000 leukocytes [<0.01%] via 8-color flow cytometry) in peripheral blood after 6 cycles of therapy.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Assessed every 2 cycles during treatment and confirmed at Cycle 6 (each cycle = 28 days)
  Proportion of participants achieving complete response (CR), partial response (PR), or partial response with lymphocytosis (PR-L) per iwCLL 2018 criteria.
Complete Response Rate (CRR) | Assessed every 2 cycles during treatment and confirmed at Cycle 6 (each cycle = 28 days)
  Proportion of participants achieving CR (normalization of blood counts, lymph nodes/spleen size, and bone marrow with <30% lymphocytes).
Progression-Free Survival (PFS) | Evaluated every 3 months post-treatment for up to 3 years.
  Time from enrollment to disease progression (per iwCLL 2018) or death from any cause.
Overall Survival (OS) | Follow-up until study completion (3 years).
  Time from enrollment to death from any cause.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From first dose to 30 days after last dose.
  Frequency and severity of adverse events graded per NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No